CLINICAL TRIAL: NCT01252264
Title: FaceBase Biorepository
Status: Completed | Type: Observational
Sponsor: Jeff Murray (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor-Investigator, Jeff Murray, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 200912764; U01DE020057 (NIH)
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Craniofacial Abnormalities; Cleft Lip; Cleft Palate
Keywords: biorepository; genetics; craniofacial; cleft lip; cleft palate
MeSH Terms: conditions — Craniofacial Abnormalities; Cleft Lip; Cleft Palate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — * A biological sample will be obtained by a blood draw. In adults, we will obtain a blood sample of 1-2 tablespoons (10-30 mL). For children, the amount will be smaller depending on their weight: 1 mL per kg to a maximum of 30 mL.
  * If a blood draw is refused, DNA can be taken from a cheek swab, spit sample or fingerstick.
  * If a participant is having surgery for a medical reason, we may request a tissue sample (for example: skin, bone, or muscle). If there were to be extra tissue, amniotic fluid, other biological samples available from a procedure performed for clinical indications, we may request a sample.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Individuals with craniofacial anomalies: Individuals who have a craniofacial anomaly (head, face, or eye disorder)
- Control Subjects: Family members of individuals with a craniofacial anomaly

SUMMARY:
The purpose of this study is to find out if there are any genetic differences between people with and without disorders of the head, face, and eye. We will create a biorepository of samples from people with and without these types of birth defects. A biorepository is a collection or "bank" of human tissue materials (such as blood or saliva) for research purposes. These samples will then be available to investigators studying these disorders.

DETAILED DESCRIPTION:
Samples from the FaceBase Biorepository and data collected from these samples will be available to investigators who are studying birth defects of the head, face, and eye. Data and samples will be deidentified prior to use by other investigators. Researchers will be allowed to use samples and medical information only after approval by the FaceBase Biorepository Data Access Committee. Once the FaceBase Biorepository Data Access Committee has established that the proposed use of the samples and clinical data meet the criteria for sound, ethical research, then the investigator will be granted permission to use a small portion of the sample and have access to clinical data stored in the computer database. Investigators who are not part of the FaceBase Biorepository Research Team will not know participant's names or other personally identifiable information.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Individual with a craniofacial anomaly or family member of an individual with a craniofacial anomaly

Exclusion Criteria:

* Non-English speaking
* Prisoners
* Minors in foster care or wards of the court

Max Age: 125 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a craniofacial anomaly and their family members.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Murray, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beaty TH, Murray JC, Marazita ML, Munger RG, Ruczinski I, Hetmanski JB, Liang KY, Wu T, Murray T, Fallin MD, Redett RA, Raymond G, Schwender H, Jin SC, Cooper ME, Dunnwald M, Mansilla MA, Leslie E, Bullard S, Lidral AC, Moreno LM, Menezes R, Vieira AR, Petrin A, Wilcox AJ, Lie RT, Jabs EW, Wu-Chou YH, Chen PK, Wang H, Ye X, Huang S, Yeow V, Chong SS, Jee SH, Shi B, Christensen K, Melbye M, Doheny KF, Pugh EW, Ling H, Castilla EE, Czeizel AE, Ma L, Field LL, Brody L, Pangilinan F, Mills JL, Molloy AM, Kirke PN, Scott JM, Arcos-Burgos M, Scott AF. A genome-wide association study of cleft lip with and without cleft palate identifies risk variants near MAFB and ABCA4. Nat Genet. 2010 Jun;42(6):525-9. doi: 10.1038/ng.580. Epub 2010 May 2. PMID 20436469
- [Background] Rahimov F, Marazita ML, Visel A, Cooper ME, Hitchler MJ, Rubini M, Domann FE, Govil M, Christensen K, Bille C, Melbye M, Jugessur A, Lie RT, Wilcox AJ, Fitzpatrick DR, Green ED, Mossey PA, Little J, Steegers-Theunissen RP, Pennacchio LA, Schutte BC, Murray JC. Disruption of an AP-2alpha binding site in an IRF6 enhancer is associated with cleft lip. Nat Genet. 2008 Nov;40(11):1341-7. doi: 10.1038/ng.242. Epub 2008 Oct 5. PMID 18836445